CLINICAL TRIAL: NCT06041451
Title: Early and Late Prognosis in Patients With Guillain-Barre Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Dengbinbin
Record Dates: First submitted 2022-12-27; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2022-12

CONDITIONS: Guillain-Barre Syndrome
Keywords: Guillain-barre syndrome; prognosis
MeSH Terms: conditions — Guillain-Barre Syndrome | interventions — Immunoglobulins, Intravenous; Methylprednisolone; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- immunoglobulin group (Experimental): This group of patients was treated with intravenous immunoglobulin(30g ivgtt qd) for 5 days
  Interventions: Drug: Intravenous Immunoglobulins, Human
- methylprednisolone group (Experimental): This group of patients was treated with methylprednisolone 500 MG Injection
  Interventions: Drug: Methylprednisolone 500 MG Injection
- control group (No Intervention): This group of patients was treated without immunoglobulin or hormone
- mixed group (Experimental): This group of patients was treated both with intravenous immunoglobulin and methylprednisolone.
  Interventions: Drug: Intravenous Immunoglobulins, Human; Drug: Methylprednisolone 500 MG Injection

INTERVENTIONS:
Drug: Intravenous Immunoglobulins, Human — patients were treated with intravenous immunoglobulin(30g ivgtt qd) for 5 days
  Arms: immunoglobulin group; mixed group
Drug: Methylprednisolone 500 MG Injection — patients were treated with methylprednisolone
  Arms: methylprednisolone group; mixed group

SUMMARY:
The goal of this observational study is to explore significant indicators to predict the early prognosis and late prognosis in patients with Guillain-Barre syndrome.

DETAILED DESCRIPTION:
This is a multicenter study(approximately three) with over 450 subjects.Clinical data were collected by consulting the patient's electronic history. The data included demographic information, blood biochemical markers, clinical characteristics and electromyography. All participants provided their written informed consent to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* patients fulfilled clinical, biological, and electrophysiology criteria for Guillain-barre syndrome.

Exclusion Criteria:

* nonidiopathic Guillain-barre syndrome and Miller Fisher syndrome

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2013-01-02 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
the severity of Guillain-barre syndrome | baseline, at 1 week, at 26 weeks
  The Guillain-barre syndrome disability score is a wide scale for the severity of Guillain-barre syndrome (0, optimal health; 1, minor symptoms, able to run; 2, able to walk unaided 10 m, unable to run; 3, able to walk 10 m across an open space with help; 4 bedridden or wheelchair users; 5, require assisted ventilation; 6, dead).The higher the score, the worse the prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China